CLINICAL TRIAL: NCT03696472
Title: Robotic-assisted Left Hemicolectomy for Left Colon Cancer With a Medial-to-lateral Approach Orientated by AMA or AMV
Brief Title: Robotic-assisted Left Hemicolectomy for Left Colon Cancer
Acronym: RALH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Li Chuan, Secretary of General Surgery, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RoboticALH
Record Dates: First submitted 2018-04-24; First posted 2018-10-04 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Robotic Surgical Procedures; Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic-assisted left colonic resection (Experimental): Standard left colonic resection assisted by Davinci Robotic
  Interventions: Procedure: robotic assisted surgery
- laparoscopic left colonic resection (Active Comparator): Standard laparoscopic left colonic resection
  Interventions: Procedure: laparoscopic

INTERVENTIONS:
Procedure: robotic assisted surgery — robotic assisted surgery was benefit to operation
  Arms: robotic-assisted left colonic resection
Procedure: laparoscopic — conventional laparoscopic surgery
  Arms: laparoscopic left colonic resection

SUMMARY:
The main goal of this study is to clarify if Robotic-assisted surgery could become the standard approach in patients undergoing left colonic resection.

Patient candidates to left colonic resection were randomly assigned to Robotic(RAL) or laparoscopic(LL) approach. The surgical staff who were not involved in the study registered 30-day postoperative morbidity. Cost-benefit analysis was based on hospital days. Long-term morbidity, quality of life, and 5-year survival have also been evaluated

DETAILED DESCRIPTION:
Robotic-assisted Left Hemicolectomy as advantages on showing the inferior mesenteric artery (IMA), protection of autonomic nerve compare to laparoscopic approach. Our experience found that operational flexibility was advantage without surgeon's position exchange.

ELIGIBILITY:
Inclusion Criteria:

Colon cancer adenocarcinoma The tumor located between the descending colon and the right 1/3 of transverse colon Tumors T3,Т4а,b N0-2 Tolerance of chemotherapy ECOG 0-2

Exclusion Criteria:

With distant metastases Tumors T1-2 Complications of tumor Women during Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
5-years overall survival rate | 5 years

SECONDARY OUTCOMES:
Short-term morbidity rate | 30 days
Anastomosis leakage rate | 6 months
Operation Time | 1 day
Blood loss during operation | 1 day
Complication incident rate of surgery | 1 day
C-reaction protein level | 7 days
Recovery time after surgery | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, China